CLINICAL TRIAL: NCT03983187
Title: Effect of Rotating Magnetic Therapy on Blood Glucose Spectrum of Type 2 Diabetic Patients With Glargine Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Majianhua (Other)
Responsible Party: Sponsor-Investigator, Majianhua, Director, Head of Endocrinology department, Clinical Professor, Nanjing First Hospital, Nanjing Medical University
Organization: Nanjing First Hospital, Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20190530-03
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Rotating Magnetic Therapy group (Experimental)
  Interventions: Device: Rotating Magnetic Therapy

INTERVENTIONS:
Device: Rotating Magnetic Therapy — Rotating Magnetic Therapy 30min/ Bid for 1 month
  Arms: Rotating Magnetic Therapy group

SUMMARY:
The aim of the study is to assess the eﬀect of Rotating Magnetic Therapy on blood glucose spectrum of type 2 diabetic patients with glargine therapy using flash glucose monitors

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate and sign informed consent prior to the study
* Patients with type 2 diabetes, who met WHO1999 diagnostic criteria, aged 18-70 years old, and were treated with insulin glargine alone and/or insulin glargine combined with oral hypoglycemic drugs, the treatment regimen was stable for more than 2 months
* Fasting blood glucose ranged from 6.1 to 13.9mmolL, and postprandial (or random) blood glucose was <22.2mmol/L.
* Subjects can and are willing to conduct flash glucose monitoring and regular diet and exercise

Exclusion Criteria:

* Patients with insulin allergy
* Patients treated with GLP-1a or DPP-4 inhibitors or multipoint subcutaneous insulin injection in the last three months
* Impaired liver and kidney function with ALT 2.5 times higher than the upper limit of normal value and serum creatinine 1.3 times higher than the upper limit of normal value
* Patients with metal foreign bodies or pacemakers
* Patients with a history of surgery in magnetic therapy site within one year
* Patients with obvious discomfort to magnetic therapy
* Patients with bleeding or bleeding tendency
* Patients with poor compliance and irregular diet and exercise
* Patients with acute complications of diabetes, such as infection, diabetic ketoacidosis, hypertonic coma and so on, and patients with stress status within four weeks
* Patients who are pregnant, breast-feeding, or intending to become pregnant
* Any other apparent conditions or associated diseases determined by the investigator: severe cardiopulmonary, endocrine, neurological, tumor, other pancreatic diseases, history of mental illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-15 (Estimated); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
the standard deviation of blood glucose | 2 weeks
  the difference of the standard deviation of blood glucose between the two groups assessed by FGM

SECONDARY OUTCOMES:
mean blood glucose | 2 weeks
  mean blood glucose between the two groups assessed by FGM
time in range | 2 weeks
  time in range assessed by FGM